CLINICAL TRIAL: NCT01249495
Title: Treatment of Chronic Legg Ulcer in Outpatient's Department and i Primary Care - Wound Size and Inflammation
Brief Title: Treatment of Chronic Leg Ulcer in Outpatient's Department and i Primary Care - Wound Size and Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); University Hospital, Aker (Other)
Responsible Party: Tone Kristin Bergersen, Oslo University hospital, Rikshospitalet, Dermatologic Department
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/736-2
Record Dates: First submitted 2010-11-25; First posted 2010-11-29 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-11

CONDITIONS: Treatment of Leg Ulcer; Sharp Debridement; Proinflammatory Cytokines
Keywords: leg ulcer; wound therapy; Pro-inflammatory interleukins
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Sharp debridement — After use of local anestetics a sharp currette is used to debride slough and nonviable tissue from the ulcer surface until a healthy tissue is seen.

SUMMARY:
The purpose of this study is to investigate the rate of wound healing using sharp debridement using curette and to compare between such intensive treatment at hospital and treatment in primary care. A correlation between change in wound size and pro-inflammatory cytokines will also be made.

DETAILED DESCRIPTION:
Subjects with chronic venous leg ulcers are treated 3 times a week in the hospital for 6 weeks with weekly sharp debridement. Wound size, pro-inflammatory cytokines, smears and photo are made weekly. The treatment countinue thereafter in primary care 3 times a week in 12 weeks. Wound size, pro-inflammatory cytokines, smears and photo are made every 14 day at the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Ulcus cruris venosoum
* AAI > 0.9
* age 18-80
* adress Oslo area
* wound size 2.5-100 cm2
* wound duration > 6 weeks.

Exclusion Criteria:

* Diabetes mellitus
* Immunosuppresion
* antibiotics < 14 days
* local antiseptic treatment < 1 week
* clinical infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-11; Primary Completion 2010-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Treatment of chronic leg ulcer in outpatient's department at hospital and in primary care - wound size and inflammation. | 01.08.10-01.08.13
  Wound size

SECONDARY OUTCOMES:
Treatment of chronic leg ulcer in outpatient's department at hospital and in primary care - wound size and inflammation. | 01.08.10-01.08.13
  Pro-inflammatory cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Tone K Bergersen, MD;PhD, Study Chair — Oslo University Hospital;Dermatologic Department
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway